CLINICAL TRIAL: NCT00643799
Title: A Randomized, Multicenter, Double-Blind, Double-Dummy Study Comparing the Efficacy and Tolerability of Once Daily Celebrex (Celecoxib) and Naproxen 500 mg Twice Daily in the 6-month Treatment of Subjects With Osteoarthritis of the Knee
Brief Title: Safety and Efficacy of Celecoxib Versus Naproxen in the 6-month Treatment of Knee Osteoarthritis
Acronym: CLOAK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3191152
Record Dates: First submitted 2008-03-18; First posted 2008-03-26 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Celecoxib; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: Celecoxib
- B (Active Comparator)
  Interventions: Drug: Naproxen
- C (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib — 200 mg oral capsule once daily for 6 months
  Arms: A
Drug: Naproxen — 500 mg oral capsule twice daily for 6 months
  Arms: B
Drug: Placebo — Matched oral placebo for 6 months
  Arms: C

SUMMARY:
To compare the safety and efficacy of celecoxib versus naproxen for the treatment of knee osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee as defined by the American College of Rheumatology criteria in a flare state at baseline visit
* Functional Capacity Classification of I-III

Exclusion Criteria:

* Inflammatory arthritis or gout/pseudo-gout with an acute flare within the past 2 years (subjects with fibrositis or fibromyalgia will not be excluded)
* Received acetaminophen within 24 hours of the baseline visit
* Acute joint trauma at index joint within the past 3 months with active symptoms
* History of gastrointestinal (GI) perforation, obstruction, or bleeding
* Diagnosed or treated for GI ulcer within 60 days prior to first dose of study medication
* Received corticosteroids or hyaluronic acid within certain timeframe before study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Actual)
Dates: Start 2004-03; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Number of responders, defined as a 20% improvement from baseline in the The Western Ontario MacMaster (WOMAC)Questionnaire Total Score | Month 6

SECONDARY OUTCOMES:
Number of health care professional contacts | Throughout study
Patient's and Physician's Satisfaction with Current Arthritis Therapy | Month 6
Change in WOMAC Total Score from baseline | Month 6
Change in WOMAC Subscales from baseline | Month 6
Response in each WOMAC Subscale | Month 6
Change in Medical Outcome Study sleep scale from baseline | Month 6
Laboratory tests | Month 6
Vital signs | Month 6
Response in VAS | Month 6
Change in Patient's and Physician's Global Assessment of Pain from baseline | Month 6
Change in visual analog scale (VAS) from baseline | Month 6
Adverse events | Throughout study
Change in Gastrointestinal (GI) Distress Scale from Week 1 | Month 6
Change in GI Distress Scale from time of discontinuation of study drug | Month 6
Receipt of prescription or over-the-counter gastroprotective agents or pain medications (off study drug) | Throughout study
Number of hospitalizations, emergency room visits, and procedures | Throughout study
Change in Work Limitation Questionnaire scale scores from baseline | Month 6
Physical examination | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- United States (44):
  - Pfizer Investigational Site, Montgomery, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tempe, Arizona
  - Pfizer Investigational Site, Buena Park, California
  - Pfizer Investigational Site, Paramount, California
  - Pfizer Investigational Site, Rancho Mirage, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Zephyrhills, Florida
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Covington, Louisiana
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, Clinton, Maryland
  - Pfizer Investigational Site, Greenbelt, Maryland
  - Pfizer Investigational Site, Hagerstown, Maryland
  - Pfizer Investigational Site, Wheaton, Maryland
  - Pfizer Investigational Site, Milford, Massachusetts
  - Pfizer Investigational Site, Lansing, Michigan
  - Pfizer Investigational Site, Flowood, Mississippi
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Beachwood, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Bethlehem, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Media, Pennsylvania
  - Pfizer Investigational Site, Warwick, Rhode Island
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, San Angelo, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191152&StudyName=Safety%20and%20Efficacy%20of%20Celecoxib%20Versus%20Naproxen%20in%20the%206-month%20Treatment%20of%20Knee%20Osteoarthritis